CLINICAL TRIAL: NCT03947840
Title: Physical Activity and Its Impact on Colon Cancer Surgery: Clinical and Histological Effects
Brief Title: Physical Activity and Its Impact on Colon Cancer Surgery
Acronym: PACOS
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Collaborators: Västerbotten County Council, Sweden (Other Government)
Responsible Party: Sponsor
Other Study IDs: PACOS
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Colon Cancer; Physical Activity
Keywords: Colon cancer; Physical activity
MeSH Terms: conditions — Colonic Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Histological samples from the tumor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Physical activity — Se their physical activity level

SUMMARY:
This is a prospective clinical study that studies how the physical activity level before operation of colon cancer affects the outcome of complication and histology.

The hypothesis is that patients who are more physical active have less postoperative complications and different histological immunological response around the tumor.

The investigators are testing the patients before the surgery with physical tests for fitness, strength and physical activity level. Questionnaires are also filled by the patients for pain, anxiety, depression and motivation for life style changes. Their body mass is analyzed with a DEXA (Dual-energy X-ray absorptiometry scan).

For one years the investigators are monitoring their activity and follow up for physical tests, DEXA and questionnaires is at 6 and 12 months.

The histology is analyzed after surgery to se if there is a different immunological response around the tumor.

ELIGIBILITY:
Inclusion Criteria:

* 18 years.
* Colon cancer which is going to surgery

Exclusion Criteria:

* Not able to do physical tests
* Severe disease that makes a risk to do tests.
* Not able to make informed consent due to psychic disease or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are going to surgery due to colon cancer.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Number of postoperative complications | 1 year
  To study if there are differences in postoperative complications in different active patients.
Rate of immunological response | 1 year
  To study if there is a difference in immunological reaction among physical active patients.

SECONDARY OUTCOMES:
Rate of recovery in physical activity | 1 year
  To study if physical active patients have a faster postoperative recovery

CONTACTS AND LOCATIONS:
Overall Officials: Karin Strigård, Principal Investigator — Umeå Universitet
Locations (1):
- Region Vasterbotten, centre of surgery, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided